CLINICAL TRIAL: NCT01732354
Title: A Prospective Study to Investigate the Consolidation Period of 12 Months Compared to 18 Months After Tenofovir Therapy With HBeAg Seroconversion in Asian Chronic Hepatitis B HBeAg-positive Patients
Brief Title: Study for Consolidation Period of Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Tainan Municipal Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IX-US-174-0206
Record Dates: First submitted 2012-11-18; First posted 2012-11-22 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis B
Keywords: Hepatitis B virus, Tenofovir
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators aim to clarify the issue of adequate duration of consolidation period of Chronic hepatitis B infection with antiviral treatment with Tenofovir which could strike a balance between durable HBeAg seroconversion and avoiding long-term inevitable serological or virological recurrence.

DETAILED DESCRIPTION:
According to practice guidelines of American Association of the Study of Liver Diseases, in patients of HBeAg-positive chronic hepatitis B, treatment should be continued until the patient has achieved HBeAg seroconversion and undetectable serum HBV DNA and completed at least 6 months of additional treatment after appearance of anti-HBe. Also several other current guidelines of anti-viral treatment of chronic hepatitis B infection suggest that nucleos (t) ide analogues treatment can be stopped following 6 to 12 months of consolidation therapy after HBeAg seroconversion. However, there is a paucity of data available about the long-term durability of Tenofovir induced HBeAg seroconversion as well as antiviral treatment associated resistance risk.

2. Primary end points: HBeAg seroconversion was defined as loss of HBeAg with concurrent appearance of HBeAb. Serological recurrence was defined as reappearance of HBeAg. Virological recurrence was defined as an increase of HBV DNA level to greater than 10,000 copies/mL after HBeAg seroconversion with previously HBV DNA levels less than 10,000 copies/mL.

3. Aims: To clarify the issue of adequate duration of consolidation period which could strike a balance between durable HBeAg seroconversion and avoiding long-term inevitable serological or virological recurrence.

4. Study design: A single-center cohort study which randomly allocating two different extended TDF treatment periods after HBeAg seroconversion - 12 months, and 18 months across patient groups. Then data will be collected about outcomes at a specific follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with chronic HBV infection (HBsAg-positivity for at least six months and HBeAg-positivity for at least three months) and serum HBV DNA levels ≥1000000 copies/ml (Cobas Amplicor HBV Monitor assay) at screening as well as serum ALT levels >1.3 times the ULN (43 IU/L) on at least two occasions in the previous 6 months and at screening.

Exclusion Criteria:

* co-infection with HCV, HDV, or HIV and treatment with (pegylated) interferon or other nucleos (t) ide analogues for less than six months before the start of Tenofovir treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 137 patients
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2013-11-20 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
HBeAg seroconversion was defined as loss of HBeAg with concurrent appearance of HBeAb. | 3 years
  We aim to clarify the issue of adequate duration of consolidation period which could strike a balance between durable HBeAg seroconversion and avoiding long-term inevitable serological or virological recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Chun-Hsiang Wang, Tainan, Taiwan